CLINICAL TRIAL: NCT01897714
Title: An Open-Label Phase I/IIa Study of the Safety and Efficacy of Melphalan-flufenamide (Melflufen) and Dexamethasone Combination for Patients With Relapsed and/or Relapsed-Refractory Multiple Myeloma
Brief Title: Safety and Efficacy of Melflufen and Dexamethasone in Relapsed and/or Relapsed-Refractory Multiple Myeloma Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated at median 46-48 months long term follow-up and mature overall survival follow-up data.
Sponsor: Oncopeptides AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: O-12-M1
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Relapsed and/or Relapsed-refractory Multiple Myeloma
MeSH Terms: interventions — melflufen; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase I: Melflufen 15 mg + Dexamethasone (Experimental): Intravenous (IV) infusion of 15 milligram (mg) melflufen on Day 1 of each 21-day treatment cycle, in combination with 40 mg dexamethasone (oral or IV) on Days 1, 8 and 15 of each 21-day treatment cycle.
  Interventions: Drug: Melflufen; Drug: Dexamethasone
- Phase I: Melflufen 25 mg + Dexamethasone (Experimental): IV infusion of 25 mg melflufen on Day 1 of each 21-day treatment cycle, in combination with 40 mg dexamethasone (oral or IV) on Days 1, 8 and 15 of each 21-day treatment cycle.
  Interventions: Drug: Melflufen; Drug: Dexamethasone
- Phase I: Melflufen 40 mg + Dexamethasone (Experimental): IV infusion of 40 mg melflufen on Day 1 of each 21-day treatment cycle, in combination with 40 mg dexamethasone (oral or IV) on Days 1, 8 and 15 of each 21-day treatment cycle.
  Interventions: Drug: Melflufen; Drug: Dexamethasone
- Phase I: Melflufen 55 mg + Dexamethasone (Experimental): IV infusion of 55 mg melflufen on Day 1 of each 21-day treatment cycle, in combination with 40 mg dexamethasone (oral or IV) on Days 1, 8 and 15 of each 21-day treatment cycle.
  Interventions: Drug: Melflufen; Drug: Dexamethasone
- Phase I + II: Melflufen 40 mg + Dexamethasone (Experimental): IV infusion of 40 mg melflufen on Day 1 of each 21-day or 28-day treatment cycles, in combination with 40 mg dexamethasone (oral or IV) on Days 1, 8 and 15 of each 21-day treatment cycles. For any patients on the 28-day treatment schedule, an additional dose of 40 mg dexamethasone was administered on Day 22 of each treatment cycle.
  Interventions: Drug: Melflufen; Drug: Dexamethasone
- Phase II: Melflufen 40 mg (Single Agent) (Experimental): IV infusion of 40 mg melflufen on Day 1 of each 28-day treatment cycle.
  Interventions: Drug: Melflufen

INTERVENTIONS:
Drug: Melflufen
Drug: Dexamethasone
  Arms: Phase I + II: Melflufen 40 mg + Dexamethasone; Phase I: Melflufen 15 mg + Dexamethasone; Phase I: Melflufen 25 mg + Dexamethasone; Phase I: Melflufen 40 mg + Dexamethasone; Phase I: Melflufen 55 mg + Dexamethasone

SUMMARY:
The study will explore escalating doses of melflufen in combination with dexamethasone in small groups of patients to find the maximum tolerated dose of melflufen. That dose will then be used to determine the efficacy and safety profile of melflufen in combination with dexamethasone in a larger group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older
2. Patient has a diagnosis of multiple myeloma with documented relapsed and/or relapsed-refractory disease
3. Patient has measurable disease defined as any of the following:

   1. Serum monoclonal protein ≥ 0.5 g/dL by protein electrophoresis
   2. ≥200 mg of monoclonal protein in the urine on 24-hour electrophoresis
   3. Serum immunoglobulin free light chain ≥10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
   4. If no monoclonal protein is detected, then ≥ 30% monoclonal bone marrow plasma cells
4. Patient has had at least 2 or more prior lines of therapy including lenalidomide and bortezomib and has demonstrated disease progression on or within 60 days of completion of the last therapy
5. Life expectancy of ≥6 months
6. Patient has an ECOG performance status ≤ 2 (Patients with lower performance status based solely on bone pain secondary to multiple myeloma will be eligible)
7. Females of childbearing potential must have a negative serum or urine pregnancy test prior to patient registration
8. Female patients of child bearing potential and non-vasectomized male patients agree to practice appropriate methods of birth control
9. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information
10. The patient has, or accepts to have, an acceptable infusion device for infusion of melflufen
11. 12 lead ECG with QtcF interval ≤ 470 msec
12. The following laboratory results must be met within 21 days of patient registration:

    * Absolute neutrophil count ≥ 1,000 cells/dL (1.0 x 109/L)
    * Platelet count ≥ 75,000 cells/dL (75 x 109/L)
    * Hemoglobin ≥ 8.0 g/dL
    * Total Bilirubin ≤ 1.5 x upper limit of normal
    * Renal function: Estimated creatinine clearance ≥ 45 ml/min or serum creatinine ≤ 2.5 mg/dL
    * AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN

Exclusion Criteria:

1. Patient has evidence of mucosal or internal bleeding and/or is platelet transfusion refractory
2. Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participation in this study
3. Known active infection requiring parenteral or oral anti-infective treatment
4. Other malignancy within the past 3 years with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, carcinoma in-situ of the cervix
5. Other ongoing anti-myeloma therapy. Patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids for symptom management and comorbid conditions. Doses of corticosteroid should be stable for at least 7 days prior to patient registration.
6. Pregnant or breast-feeding females
7. Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation
8. Known HIV or hepatitis B or C viral infection
9. Patient has concurrent symptomatic amyloidosis or plasma cell leukemia
10. POEMS syndrome
11. Previous cytotoxic therapies, including cytotoxic investigational agents, for multiple myeloma within 3 weeks (6 weeks for nitrosoureas) prior to start of study treatment. Biologic, novel therapy (including investigational agents in this class) or corticosteroids within 2 weeks prior to patient registration. Patient has side effects of the previous therapy > grade 1 or previous baseline.
12. Prior peripheral stem cell transplant within 12 weeks of patient registration
13. Radiotherapy within 21 days prior to Cycle 1 Day 1. However, if the radiation portal covered ≤ 5% of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy
14. Known intolerance to steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Richardson, MD, Study Director — Dana Farber Cancer Institute, Boston MA, USA; Johan Harmenberg, MD, Study Director — Oncopeptides AB, Stockholm, Sweden
Locations (7):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Universtity of North Carolina, Chapel Hill, North Carolina
- Vejle Hospital, Vejle, Denmark
- Turin Hospital Myeloma Unit, Turin, Italy
- Erasmus University Medical Center, Rotterdam, Netherlands
- Sahlgrenska Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Richardson PG, Bringhen S, Voorhees P, Plesner T, Mellqvist UH, Reeves B, Paba-Prada C, Zubair H, Byrne C, Chauhan D, Anderson K, Nordstrom E, Harmenberg J, Palumbo A, Sonneveld P. Melflufen plus dexamethasone in relapsed and refractory multiple myeloma (O-12-M1): a multicentre, international, open-label, phase 1-2 study. Lancet Haematol. 2020 May;7(5):e395-e407. doi: 10.1016/S2352-3026(20)30044-2. Epub 2020 Mar 23. PMID 32213344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, Phase I/IIa study conducted at 7 study centers in 5 countries in patients with relapsed and/or relapsed-refractory Multiple Myeloma (MM). Overall, 75 patients (23 during Phase I and 52 additional patients during Phase II) were enrolled. The study results are presented until the end of trial (EOT) date of 29 October 2019.
Pre-assignment Details: The study was conducted in 2 parts: Phase I (dose escalation) and Phase II (maximum tolerated dose [MTD]). During Phase I, the standard 3 + 3 design was followed with 3 to 6 patients tested at each dose level, depending on the dose limiting toxicity (DLT) observed. During Phase II, patients were treated at the MTD determined in Phase I.
Groups:
- Phase I: Melflufen 15 mg + Dexamethasone: Patients were treated with 15 milligram (mg) melflufen as intravenous (IV) infusion on Day 1 and 40 mg dexamethasone oral tablet or IV infusion on Days 1, 8 and 15 of each 21-day treatment cycle. Patients could continue receiving treatment for up to 8 cycles or until they experienced unacceptable toxicity, disease progression, withdrew consent, and/or the study drug was discontinued at the discretion of the Investigator.
- Phase I: Melflufen 25 mg + Dexamethasone: Patients were treated with 25 mg melflufen as IV infusion on Day 1 and 40 mg dexamethasone oral tablet or IV infusion on Days 1, 8 and 15 of each 21-day treatment cycle. Patients could continue receiving treatment for up to 8 cycles or until they experienced unacceptable toxicity, disease progression, withdrew consent, and/or the study drug was discontinued at the discretion of the Investigator.
- Phase I: Melflufen 40 mg + Dexamethasone: Patients were treated with 40 mg melflufen as IV infusion on Day 1 and 40 mg dexamethasone oral tablet or IV infusion on Days 1, 8 and 15 of each 21-day treatment cycle. Patients could continue receiving treatment for up to 8 cycles or until they experienced unacceptable toxicity, disease progression, withdrew consent, and/or the study drug was discontinued at the discretion of the Investigator.
- Phase I: Melflufen 55 mg + Dexamethasone: Patients were treated with 55 mg melflufen as IV infusion on Day 1 and 40 mg dexamethasone oral tablet or IV infusion on Days 1, 8 and 15 of each 21-day treatment cycle. Patients could continue receiving treatment for up to 8 cycles or until they experienced unacceptable toxicity, disease progression, withdrew consent, and/or the study drug was discontinued at the discretion of the Investigator.
- Phase I + II: Melflufen 40 mg + Dexamethasone: Patients were treated with 40 mg melflufen as IV infusion on Day 1 and 40 mg dexamethasone oral tablet or IV infusion on Days 1, 8 and 15 of each 21-day or 28-day treatment cycle. Patients could continue receiving treatment for up to 8 cycles or until they experienced unacceptable toxicity, disease progression, withdrew consent, and/or the study drug was discontinued at the discretion of the Investigator. In Protocol amendment 4, the cycle of melflufen was increased from 21 to 28 days. For any patients on the 28-day treatment schedule, an additional dose of 40 mg dexamethasone was administered on Day 22 of each cycle.
- Phase II: Melflufen 40 mg (Single Agent): Patients were treated with 40 mg melflufen as IV infusion on Day 1 of each 28-day treatment cycle. Dexamethasone was not administered as an antitumor compound. However, all patients were treated with 8 mg dexamethasone as an antiemetic on Days 1 and 2, and an optional 4 mg dexamethasone as an antiemetic on Days 3 and 4 of the same 28-day cycle, unless the Investigator decided to switch a patient to a combination regimen. Patients could continue receiving treatment for up to 8 cycles or until they experienced unacceptable toxicity, disease progression, withdrew consent, and/or the study drug was discontinued at the discretion of the Investigator.
Period: Phase I (Dose Escalation)
Arm/Group | Phase I: Melflufen 15 mg + Dexamethasone | Phase I: Melflufen 25 mg + Dexamethasone | Phase I: Melflufen 40 mg + Dexamethasone | Phase I: Melflufen 55 mg + Dexamethasone | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Started | 4 | 7 | 6 | 6 | 0 | 0
Completed (Completed 8 cycles or more of study drug.) | 1 | 0 | 1 | 0 | 0 | 0
Not Completed | 3 | 7 | 5 | 6 | 0 | 0
Not completed — Disease progression | 3 | 5 | 1 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 4 | 3 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0
Period: Phase II (MTD)
Arm/Group | Phase I: Melflufen 15 mg + Dexamethasone | Phase I: Melflufen 25 mg + Dexamethasone | Phase I: Melflufen 40 mg + Dexamethasone | Phase I: Melflufen 55 mg + Dexamethasone | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Started | 0 | 0 | 0 | 0 | 45 (6 patients were entered from the Phase I: Melflufen 40 mg + Dexamethasone arm.) | 13
Completed | 0 | 0 | 0 | 0 | 15 | 2
Not Completed | 0 | 0 | 0 | 0 | 30 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 25 | 10
Not completed — Study terminated with patient alive | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all patients who received at least 1 dose, or part thereof, of study drug.
Groups:
- Phase I: Melflufen 15 mg + Dexamethasone: Patients were treated with 15 mg melflufen as IV infusion on Day 1 and 40 mg dexamethasone oral tablet or IV infusion on Days 1, 8 and 15 of each 21-day treatment cycle. Patients could continue receiving treatment for up to 8 cycles or until they experienced unacceptable toxicity, disease progression, withdrew consent, and/or the study drug was discontinued at the discretion of the Investigator.
- Total: Total of all reporting groups
Arm/Group | Phase I: Melflufen 15 mg + Dexamethasone | Phase I: Melflufen 25 mg + Dexamethasone | Phase I: Melflufen 40 mg + Dexamethasone | Phase I: Melflufen 55 mg + Dexamethasone | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent) | Total
Number analyzed (Participants) | 4 | 7 | 6 | 6 | 45 | 13 | 81
Age, Categorical [Count of Participants; unit: Participants] — Population: 6 patients from the Phase I: Melflufen 40 mg + Dexamethasone arm were transferred to Phase I + II: Melflufen 40 mg + Dexamethasone arm. All arms for the baseline analysis were not mutually exclusive (mutually exclusive patients = 75).
  Participants
    Phase I: number analyzed (Participants) | 4 | 7 | 6 | 6 | 0 | 0 | 23
    Phase I: <=18 years | 0 | 0 | 0 | 0 |  |  | 0
    Phase I: Between 18 and 65 years | 1 | 3 | 3 | 2 |  |  | 9
    Phase I: >=65 years | 3 | 4 | 3 | 4 |  |  | 14
    Phase II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 13 | 58
    Phase II: <=18 years |  |  |  |  | 0 | 0 | 0
    Phase II: Between 18 and 65 years |  |  |  |  | 20 | 8 | 28
    Phase II: >=65 years |  |  |  |  | 25 | 5 | 30
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 6 patients from the Phase I: Melflufen 40 mg + Dexamethasone arm were transferred to Phase I + II: Melflufen 40 mg + Dexamethasone arm. All arms for the baseline analysis were not mutually exclusive (mutually exclusive patients = 75).
  Participants
    Phase I: number analyzed (Participants) | 4 | 7 | 6 | 6 | 0 | 0 | 23
    Phase I: Female | 2 | 4 | 2 | 3 |  |  | 11
    Phase I: Male | 2 | 3 | 4 | 3 |  |  | 12
    Phase II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 13 | 58
    Phase II: Female |  |  |  |  | 15 | 5 | 20
    Phase II: Male |  |  |  |  | 30 | 8 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 6 patients from the Phase I: Melflufen 40 mg + Dexamethasone arm were transferred to Phase I + II: Melflufen 40 mg + Dexamethasone arm. All arms for the baseline analysis were not mutually exclusive (mutually exclusive patients = 75).
  Participants
    Phase I: number analyzed (Participants) | 4 | 7 | 6 | 6 | 0 | 0 | 23
    Phase I: Black or African American | 1 | 1 | 0 | 0 |  |  | 2
    Phase I: Caucasian | 3 | 6 | 6 | 6 |  |  | 21
    Phase I: Not collected as per local laws | 0 | 0 | 0 | 0 |  |  | 0
    Phase II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 13 | 58
    Phase II: Black or African American |  |  |  |  | 3 | 3 | 6
    Phase II: Caucasian |  |  |  |  | 41 | 10 | 51
    Phase II: Not collected as per local laws |  |  |  |  | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 6 patients from the Phase I: Melflufen 40 mg + Dexamethasone arm were transferred to Phase I + II: Melflufen 40 mg + Dexamethasone arm. All arms for the baseline analysis were not mutually exclusive (mutually exclusive patients = 75).
  Participants
    Phase I: number analyzed (Participants) | 4 | 7 | 6 | 6 | 0 | 0 | 23
    Phase I: Hispanic or Latino | 0 | 1 | 0 | 0 |  |  | 1
    Phase I: Not Hispanic or Latino | 4 | 6 | 5 | 5 |  |  | 20
    Phase I: Not collected as per local laws | 0 | 0 | 1 | 1 |  |  | 2
    Phase II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 13 | 58
    Phase II: Hispanic or Latino |  |  |  |  | 1 | 0 | 1
    Phase II: Not Hispanic or Latino |  |  |  |  | 37 | 12 | 49
    Phase II: Not collected as per local laws |  |  |  |  | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Achieved Best Overall Disease Response
Description: The best overall disease response on treatment including stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR), stable disease (SD) or progressive disease (PD) were evaluated. Starting on completion of Cycle 2, response was assessed according to International Myeloma Working Group (IMWG) criteria based on Investigator's assessment for all patients at every cycle during treatment period. PD was defined as increase of ≥25% from lowest response value in any 1 of the following: serum M-component (absolute increase must be ≥0.5 gram/deciliter) and/or urine M-component (absolute increase must be ≥200 mg/24 hr); development of new bone lesions or soft tissue plasmacytomas or increase in size of existing bone lesions or soft tissue plasmacytomas or development of hypercalcemia that could be attributed solely to plasma cell proliferative disorder. SD was defined as not meeting criteria for CR, VGPR, PR or PD.
Time Frame: Baseline (Cycle 1 Day 1) and every cycle from Cycle 2 onwards until confirmed disease progression. Assessed until EOT date of 29 October 2019; up to a maximum of approximately 76 months.
Population: For Phase I arms: The Safety Analysis Set included all patients who received at least 1 dose, or part thereof, of study drug.
  For Phase II arms: Modified Intent-to-Treat (mITT) Analysis Set included all patients considered to be valid for Safety Analysis Set and who received at least 1 dose of study drug at the MTD as initial dose.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Phase I: Melflufen 15 mg + Dexamethasone | Phase I: Melflufen 25 mg + Dexamethasone | Phase I: Melflufen 40 mg + Dexamethasone | Phase I: Melflufen 55 mg + Dexamethasone | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 4 | 7 | 6 | 6 | 45 | 13
percentage of patients
  sCR | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 24.7]
  CR | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 24.7]
  VGPR | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 11.1 [3.7 to 24.1] | 0.0 [0.0 to 24.7]
  PR | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 50.0 [11.8 to 88.2] | 0.0 [0.0 to 45.9] | 20.0 [9.6 to 34.6] | 7.7 [0.2 to 36.0]
  MR | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 17.8 [8.0 to 32.1] | 15.4 [1.9 to 45.4]
  SD | 75.0 [19.4 to 99.4] | 42.9 [9.9 to 81.6] | 16.7 [0.4 to 64.1] | 66.7 [22.3 to 95.7] | 26.7 [14.6 to 41.9] | 69.2 [38.6 to 90.9]
  PD | 25.0 [0.6 to 80.6] | 57.1 [18.4 to 90.1] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 15.6 [6.5 to 29.5] | 7.7 [0.2 to 36.0]
  Missing | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 8.9 [2.5 to 21.2] | 0.0 [0.0 to 24.7]
  sCR + CR | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 24.7]
  sCR + CR + VGPR | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 11.1 [3.7 to 24.1] | 0.0 [0.0 to 24.7]

2. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as percentage of patients with an overall response (OR), defined as first occurrence of confirmed disease response including PR or better (i.e, PR, VGPR, CR or sCR). Starting on completion of Cycle 2, response was assessed according to IMWG criteria based on Investigator's assessment for all patients at every cycle during treatment period. VGPR was defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum plus urine M-protein level <100 mg/24hr and >90% decrease in difference between involved and uninvolved free light chain (FLC) levels (only in FLC diseased patients). CR was defined as negative immunofixation on serum and urine, loss of any soft tissue plasmacytomas, <5% plasma cells in bone marrow and normal FLC ratio of 0.26 to 1.65 (only in FLC diseased patients). sCR was defined as CR plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or 2 to 4 color flow cytometry.
Time Frame: Baseline and every cycle from Cycle 2 onwards until confirmed disease progression. Assessed until EOT date of 29 October 2019; up to a maximum of approximately 76 months.
Population: For Phase I arms: The Safety Analysis Set included all patients who received at least 1 dose, or part thereof, of study drug.
  For Phase II arms: The mITT Analysis Set included all patients considered to be valid for the Safety Analysis Set and who received at least 1 dose of study drug at the MTD as the initial dose.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Phase I: Melflufen 15 mg + Dexamethasone | Phase I: Melflufen 25 mg + Dexamethasone | Phase I: Melflufen 40 mg + Dexamethasone | Phase I: Melflufen 55 mg + Dexamethasone | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 4 | 7 | 6 | 6 | 45 | 13
percentage of patients | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 66.7 [22.3 to 95.7] | 16.7 [0.4 to 64.1] | 31.1 [18.2 to 46.6] | 7.7 [0.2 to 36.0]

3. Primary Outcome: Clinical Benefit Response Rate (CBRR)
Description: The CBRR was defined as the percentage of patients with a clinical benefit response (CBR), defined as the first occurrence of confirmed disease response including MR or better (i.e, MR, PR, VGPR, CR, or sCR). Starting on completion of Cycle 2, response was assessed according to the IMWG criteria based on the Investigator's assessment for all patients at every cycle during the treatment period. MR was defined as ≥25% but <49% reduction of serum M-protein and reduction in 24 hour urine M-protein by 50 to 89%, which still exceeds 200 mg/24 hours. In addition to above; if present at baseline, 25 to 49% reduction in the size of soft tissue plasmacytomas is also required. No increase in size or number of lytic bone lesions (development of compression fractures does not exclude response). PR was defined as 50% reduction of serum M-protein and reduction in 24 hour urinary M-protein by ≥90% or to <200 mg/24 hour.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Phase I: Melflufen 15 mg + Dexamethasone | Phase I: Melflufen 25 mg + Dexamethasone | Phase I: Melflufen 40 mg + Dexamethasone | Phase I: Melflufen 55 mg + Dexamethasone | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 4 | 7 | 6 | 6 | 45 | 13
percentage of patients | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 41.0] | 66.7 [22.3 to 95.7] | 16.7 [0.4 to 64.1] | 48.9 [33.7 to 64.2] | 23.1 [5.0 to 53.8]

4. Secondary Outcome: Duration of Disease Response (DOR)
Description: The DOR to treatment was defined as time from first response (PR or better) to disease progression or death, or date of last evaluable disease response assessment for those who had not progressed or died. DOR was estimated using Kaplan-Meier statistics.
Time Frame: as for outcome 2
Population: The mITT Analysis Set included all patients considered to be valid for the Safety Analysis Set and who received at least 1 dose of study drug at the MTD as the initial dose. Only patients who had achieved at least PR were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 14 | 1
months | 8.4 [4.6 to 11.1] | 7.2 [NA to NA] — The confidence interval could not be determined as only 1 patient was analysed.

5. Secondary Outcome: Time to Disease Response in Patients Who Achieved OR and CBR
Description: Time to first OR was defined as the time from the date of the first dose of study drug (overall reference start date) to the date of the first occurrence of PR or better (first of 2 consecutive assessments-confirmed response). Time to first CBR was defined as the time from the date of the first dose of study drug (overall reference start date) to the date of the first occurrence of MR or better (first of 2 consecutive assessments-confirmed response). Time to disease response was estimated using Kaplan-Meier statistics.
Time Frame: as for outcome 2
Population: The mITT Analysis Set included all patients considered to be valid for the Safety Analysis Set and who received at least 1 dose of study drug at the MTD as the initial dose. Only patients who had achieved OR and CBR were evaluated, for each respective time to response parameter.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 22 | 3
months
  OR: number analyzed (Participants) | 14 | 1
  OR | 2.8 [1.6 to 4.7] | 6.7 [NA to NA] — The confidence interval could not be determined as only 1 patient was analysed.
  CBR | 2.4 [1.4 to 3.0] | 2.8 [2.8 to 6.1]

6. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from the date of the first dose of study drug (overall reference start date) to the date of the first occurrence of evaluable PD. Time to disease progression was estimated using Kaplan-Meier statistics.
Time Frame: as for outcome 2
Population: The mITT Analysis Set included all patients considered to be valid for the Safety Analysis Set and who received at least 1 dose of study drug at the MTD as the initial dose.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 45 | 13
months | 6.5 [3.7 to 9.3] | 4.4 [2.8 to 12.2]

7. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: The PFS was defined as the time from the date of the first dose of melflufen (overall reference start date) to the date of the first occurrence of any disease response assessment available for PD or death. The PFS was estimated using Kaplan-Meier statistics.
Time Frame: as for outcome 2
Population: The mITT Analysis Set included all patients considered to be valid for the Safety Analysis Set and who received at least 1 dose of study drug at the MTD as the initial dose. Only patients who had information about PFS at the time of EOT (29 October 2019) were reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 45 | 13
months | 5.7 [3.7 to 9.2] | 4.4 [2.8 to 7.6]

8. Secondary Outcome: Median Overall Survival (OS)
Description: The OS was defined as the time from the date of the first dose of melflufen (overall reference start date) to death. The OS was estimated using Kaplan-Meier statistics.
Time Frame: From baseline until death. Assessed until EOT date of 29 October 2019; up to a maximum of approximately 76 months.
Population: The mITT Analysis Set included all patients considered to be valid for the Safety Analysis Set and who received at least 1 dose of study drug at the MTD as the initial dose. Only patients who had information about OS at the time of EOT(29 October 2019) were reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 45 | 13
months | 20.7 [11.8 to 41.3] | 15.5 [4.9 to 23.4]

9. Secondary Outcome: Time to First Subsequent Treatment
Description: Time to first subsequent treatment start was defined as the time from the date of the actual end of treatment to the date of the first subsequent treatment. Time to first subsequent treatment was estimated using Kaplan-Meier statistics.
Time Frame: From baseline until start of first subsequent treatment. Assessed until EOT date of 29 October 2019; up to a maximum of approximately 76 months.
Population: The mITT Analysis Set included all patients considered to be valid for the Safety Analysis Set and who received at least 1 dose of study drug at the MTD as the initial dose. Only patients who had information about first subsequent treatment at the time of EOT (29 October 2019) were reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 45 | 13
months | 10.5 [7.9 to 12.2] | 10.7 [5.3 to NA] — Upper limit of confidence could not be calculated as it was not reached.

10. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a study patient administered an investigational product and that does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was defined as any AE, occurring at any dose, that met any one or more of the following criteria: is fatal or immediately life-threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; is medically significant; requires inpatient hospitalization or prolongation of existing hospitalization; or other important medical event. TEAEs were defined as AEs that started or worsened on or after the first dose of study drug (overall reference start date) up to and including the actual EOT date. TESAEs = Treatment emergent serious adverse events.
Time Frame: From the first dose of study drug up to and including the actual EOT date of 29 October 2019; up to a maximum of approximately 76 months.
Population: The Safety Analysis Set included all patients who received at least 1 dose, or part thereof, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Melflufen 15 mg + Dexamethasone | Phase I: Melflufen 25 mg + Dexamethasone | Phase I: Melflufen 40 mg + Dexamethasone | Phase I: Melflufen 55 mg + Dexamethasone | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
Number analyzed (Participants) | 4 | 7 | 6 | 6 | 45 | 13
Participants
  TEAEs (including both serious and non-serious AEs) | 4 | 7 | 6 | 6 | 45 | 13
  TEAEs leading to death | 0 | 1 | 0 | 0 | 3 | 0
  TESAEs | 3 | 4 | 2 | 4 | 17 | 9
  DLT TEAEs: number analyzed (Participants) | 4 | 7 | 6 | 6 | 0 | 0
  DLT TEAEs | 0 | 0 | 0 | 4 |  |
  TEAEs related to melflufen and/or dexamethasone | 4 | 7 | 6 | 6 | 45 | 13
  TESAEs related to melflufen and/or dexamethasone | 3 | 4 | 2 | 4 | 17 | 9

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to and including the actual EOT date of 29 October 2019; up to a maximum of approximately 76 months.
Description: The Safety Analysis Set included all patients who received at least 1 dose, or part thereof, of study drug.
Arm/Group | Phase I: Melflufen 15 mg + Dexamethasone | Phase I: Melflufen 25 mg + Dexamethasone | Phase I: Melflufen 40 mg + Dexamethasone | Phase I: Melflufen 55 mg + Dexamethasone | Phase I + II: Melflufen 40 mg + Dexamethasone | Phase II: Melflufen 40 mg (Single Agent)
All-Cause Mortality (participants affected / at risk) | 3/4 | 5/7 | 2/6 | 5/6 | 30/45 | 10/13
Serious Adverse Events (participants affected / at risk) | 3/4 | 4/7 | 2/6 | 4/6 | 17/45 | 9/13
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 6/6 | 6/6 | 45/45 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Melflufen 15 mg + Dexamethasone (N=4) | Phase I: Melflufen 25 mg + Dexamethasone (N=7) | Phase I: Melflufen 40 mg + Dexamethasone (N=6) | Phase I: Melflufen 55 mg + Dexamethasone (N=6) | Phase I + II: Melflufen 40 mg + Dexamethasone (N=45) | Phase II: Melflufen 40 mg (Single Agent) (N=13)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (10)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Melflufen 15 mg + Dexamethasone (N=4) | Phase I: Melflufen 25 mg + Dexamethasone (N=7) | Phase I: Melflufen 40 mg + Dexamethasone (N=6) | Phase I: Melflufen 55 mg + Dexamethasone (N=6) | Phase I + II: Melflufen 40 mg + Dexamethasone (N=45) | Phase II: Melflufen 40 mg (Single Agent) (N=13)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 6 (9) | 4 (26) | 5 (35) | 33 (154) | 9 (30)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (7) | 3 (12) | 6 (26) | 31 (115) | 9 (25)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (5) | 2 (4) | 3 (6) | 29 (96) | 5 (14)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (6) | 4 (5) | 12 (14) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 7 (8) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (5) | 9 (10) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (5) | 3 (7) | 2 (2) | 13 (20) | 4 (4)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 16 (19) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 6 (8) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 14 (46) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 6 (9) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (8) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 5 (6) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 3 (5) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 6 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (11) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (8) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 6 (8) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucous membrane disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibrin d dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin B12 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (13) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve disease mixed (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune system disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Study is terminated and long-term follow-up ended due to Sponsor decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT01897714/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT01897714/SAP_001.pdf